CLINICAL TRIAL: NCT03557632
Title: University of Houston Drug Abuse Research Development Program II
Acronym: UHDARDP-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Luis R. Torres, PhD, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R24DA019798-08 REVISED; 5R24DA019798 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-06-15 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Heroin Dependence
Keywords: Opioid Dependence; Injection Drug Use; Hispanics; Mexican Americans; Virtual Reality Cue Exposure
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The proposed study will use a between-groups, randomized controlled experimental design to test the effects of Virtual Reality Cue Exposure Therapy (VRCET) compared to Relapse Prevention Drug Education (RPDE) on self-reported drug craving, physiological reactivity (i.e., Galvanic Skin Conductance [GSC] and heart rate [HR]), craving coping skills, and drug use among Mexican American IDUs and NIDUs with heroin as their primary drug of choice (see design below). All participants who are former IDU will not be randomized and will complete the VRCET protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT:Virtual Reality Cue Exposure Therapy (VRCET) (Experimental): Virtual Reality Cue Exposure Therapy (VRCET) - Active Intervention - comprised of exposure to VR based heroin cues, such as heroin use paraphernalia and scenes of people using injection heroin or snorting heroin. Exposure will be supplemented by the use of a standardized CBT based skills coping protocol teaching relapse prevention skills such as urge surfing, thought stopping and reframing. Lab based reactivity will be measured by self-reported craving on a scale from 0 (none) to 100 (highest ever), heart rate, galvanic skin response, and muscle tension. Secondary outcome measures are number of times of self-reported drug use in vivo as recorded by a cell phone app based Ecological Momentary Assessment Device (EMA).
  Interventions: Behavioral: Virtual Reality Cue Exposure Therapy
- Control: Relapse Prevention Drug Education (Active Comparator): Relapse Prevention Drug Education (RPDE) is our Active Comparator. Comprised of watching a series of videos on the health risks of heroin use as well as information about relapse prevention. Lab based reactivity will be measured by self-reported craving on a scale from 0 (none) to 100 (highest ever), heart rate, galvanic skin response, and muscle tension. Secondary outcome measures are number of times of self-reported drug use in vivo as recorded by a cell phone app based Ecological Momentary Assessment Device (EMA).
  Interventions: Behavioral: Relapse Prevention Drug Education

INTERVENTIONS:
Behavioral: Virtual Reality Cue Exposure Therapy — As above.
  Arms: TREATMENT:Virtual Reality Cue Exposure Therapy (VRCET)
Behavioral: Relapse Prevention Drug Education — As above.
  Arms: Control: Relapse Prevention Drug Education

SUMMARY:
The study is examining the impact of a Virtual Reality Cue Exposure Therapy intervention on heroin cravings compared to Relapse Prevention Drug Education.

DETAILED DESCRIPTION:
Injection Drug Use (IDU) is a chronic, relapsing condition with grave individual and public health consequences.19-21 A majority (53%) of all past-year IDUs prefer heroin, as do 39% of single-drug injectors, second only to Methamphetamine.22,23 Non-injection heroin use (NIDU) is increasing, due to growing awareness of IDU risks, particularly HIV/AIDS;21,24-26 increased purity of street heroin;27-29 greater regulation of other opiates;30,31 and opioid abusers switching to heroin for its lower cost.32 Many NIDUs transition to IDU, incurring greater risks.2,21,33,34 Drug cravings are intense urges to use drugs35,36 and they contribute to drug use37, relapse38, and transitioning from NIDU to IDU.39 Cravings are triggered by environmental factors and due to the significance of craving in drug use and relapse they will be part of the proposed criteria for DSM5.40,41

HIV, Hepatitis C (HCV), and Sexually-Transmitted Infections (STIs) continue to be associated with both IDU and NIDU.33,42-44 Hispanics are over-represented among both IDU and NIDU heroin users.21,23,45,46 Mexican American IDUs have very low rates of HIV.10,47 However, their HCV rates are very high and continue to increase, further compromising their health.10,48,49 They also have elevated rates of high-risk sex behaviors 33,50 and they are less likely to decrease these high-risk sex behaviors than they are to decrease their injection- behavior risks, especially as they age.10,51 Furthermore, HIV/HCV/STI prevention interventions can lead to fatigue52-54 so they must continue to be delivered to at-risk populations across all relevant settings. Young Texans ages 15-24 are becoming HIV infected at high rates, with Hispanics disproportionately impacted and diagnosed later: 42% of infected Texan Hispanics receive an HIV-positive and an AIDS diagnosis within the same year, compared to 32% of Anglos and 31% of Blacks.55 Thus, early detection of high-risk Hispanics is vital, making this proposal timely and critical.

Greatly needed are novel interventions that address drug cravings (DCs), take into account environmental context, and incorporate HIV/HCV prevention components. Developing these interventions and adapting them to the many diverse at-risk populations, however, can be costly and challenging. Cue exposure therapy (CET)56,57 may be a viable approach. CET is a promising intervention that can decrease DCs by repeatedly exposing an individual to a craving inducing stimulus (e.g., a shooting gallery scenario) while simultaneously preventing the conditioned behavioral response (e.g., drug use). The individual can be trained in vitro (in the lab) to use coping skills in direct response to activated cravings, then use these skills in vivo (in the natural environment). A challenge associated with CET, for both ethical and logistical reasons, is the ability to expose individuals to realistic simulated cues of the natural environment in a secure laboratory or therapeutic setting. Virtual Reality (VR) is an innovative, cutting-edge tool that can enable researchers to overcome these obstacles. VR scenarios integrate elements from the individual's various contexts-culture, neighborhood, family, networks, and individual characteristics-into the clinical or lab setting, and provide complex multi-sensory cues through an immersive human-computer interaction.58

The public health significance of this primary project is high. Drug use in general and injection drug use (IDU) in particular are serious public health concerns, as are the rates of HCV and STIs in IDUs. Interventions that decrease craving, increase coping skills, and incorporate HIV/HCV/STI prevention components can be critical tools in treating drug use disorders and their serious health consequences. In addition, it is critical to train diverse researchers who possess intimate knowledge of the populations impacted by drug use and who understand the cultural and contextual elements of those populations, to conduct this innovative research.

The specific research hypotheses and objectives are as follows:

1. Refine and develop a Virtual Reality Heroin Scenario (VRHS) using qualitative data (i.e., photos and descriptions of heroin using sites and contexts) from our current UHDARDP's Primary Project.
2. Measure the effects of exposure to virtual reality heroin cues on craving and physiological reactivity.

   Hypothesis 1a: VR cues will increase subjective heroin craving and physiological reactivity.

   Hypothesis 1b: Heroin craving and physiological reactivity will decrease as a result of repeated exposure to virtual cues.
3. Compare Virtual Reality-Based Cue Exposure Therapy (VRCET) and Relapse Prevention Drug Education (RPDE) on extinction of heroin craving and physiological reactivity across cue trials.

   Hypothesis 2: VRCET will attenuate cue-elicited subjective heroin craving and physiological reactivity relative to RPDE.
4. Examine the in vivo effects of VRCET on heroin craving, craving coping skills, and actual heroin use, compared to RPDE.

   Hypothesis 3: VRCET will lead to a decrease in heroin craving, an increase in craving coping skills use, and decreased heroin use, in the natural environment, compared to RPDE.
5. Deliver an HIV/HCV prevention intervention to this high-risk population. Hypothesis 4: The prevention intervention will increase prevention knowledge and intention to use the skills learned.
6. Determine if medication assisted therapies, such as methadone or buprenorphine, have an impact on cue reactivity for former heroin IDU when immersed in the virtual environments, as compared to current users.

Hypothesis 5: Participants on medication assisted therapies will exhibit lower levels of cue reactivity within the VR environment than participants who are currently still using heroin.

ELIGIBILITY:
Inclusion Criteria:

* Injection or Non-Injection heroin user, 3 or more years of heroin use, Hispanic/Latino

Exclusion Criteria:

* Non heroin user, non-Hispanic/Latino, younger than 18 or older than 64, treated with any medications having a potential effect on heroin craving, mood, or heroin cessation medications in the past 30 days; use of other prescription and non-prescription drugs that may affect participation; Fear of closed spaces or inability to wear VR goggles; Visual problems that effect viewing VR materials; History of seizures or seizure disorders; History of serious self-reported health problems; and women who are pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported reactivity to cues | 3 hours (6 blocks of 3 minutes with time in between each block); this is done in two consecutive weeks.
  Self-reported craving on a scale from 0 (none) to 100 (highest ever)
Lab-based reactivity to cues | 3 hours (6 blocks of 3 minutes with time in between each block); this is done in two consecutive weeks. These are monitored continuously every 10th of a second.
  Heart rate (ECG) assessed in beats per minute using a Bioradio Wireless Physiology (see https://glneurotech.com/bioradio/psychophysiology-equipment/).
Lab-based reactivity to cues | 3 hours (6 blocks of 3 minutes with time in between each block); this is done in two consecutive weeks. These are monitored continuously every 10th of a second.
  Galvanic skin response (GSR) assessed using a Bioradio Wireless Physiology (see https://glneurotech.com/bioradio/psychophysiology-equipment/).
Lab-based reactivity to cues | 3 hours (6 blocks of 3 minutes with time in between each block); this is done in two consecutive weeks. These are monitored continuously every 10th of a second.
  Changes in muscle tension (EMG) assessed using a Bioradio Wireless Physiology (see https://glneurotech.com/bioradio/psychophysiology-equipment/).

SECONDARY OUTCOMES:
Number of times of self-reported drug use in vivo during the week between lab sessions. | Continuously during the 4 weeks
  As recorded by a cell phone app based Ecological Momentary Assessment Device (EMA)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston Virtual Reality Clinical Research Lab, Houston, Texas, United States